CLINICAL TRIAL: NCT03048929
Title: Effects of Inflammation on Neural Mechanisms of Threat Sensitivity in Posttraumatic Stress Disorder
Brief Title: Inflammation and Threat Sensitivity in PTSD
Acronym: K01
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-18367; K01MH109871 (NIH)
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Typhoid Vi Polysaccharide Vaccine (Active Comparator): Patients will receive one intramuscular 0.5 mL injection of Typhoid Vi Polysaccharide Vaccine containing 0.025 mg purified Vi polysaccharide.
  Interventions: Biological: Typhoid Vi Polysaccharide Vaccine
- Placebo (Placebo Comparator): Patients will receive one intramuscular 0.5 mL injection of saline placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Typhoid Vi Polysaccharide Vaccine — Salmonella typhi capsular polysaccharide vaccine (Typhoid Vi Polysaccharide Vaccine): Each dose of 0.5ml Salmonella typhi capsular polysaccharide vaccine (Sanofi Pasteur, SA) is formulated to contain 25μg of purified Vi polysaccharide in a colorless isotonic phosphate buffered saline (pH 7±0.3), 4.150mg of sodium chloride, 0.065mg of disodium phosphate, 0.023mg of monosodium phosphate and 0.5ml of sterile water for injection. It is indicated for use by humans aged 2 years and older for protection against typhoid fever.
  Arms: Typhoid Vi Polysaccharide Vaccine
Biological: Placebo — The placebo injection will consist of 0.5mL of saline.
  Arms: Placebo

SUMMARY:
The overall goals of this study are to examine the relationship between chronic inflammation and threat and reward sensitivity, and to determine the effects of acute inflammation on threat sensitivity, in individuals with and without moderate to severe PTSD symptoms. The investigators will first conduct an observational study to examine the relationship between chronic inflammation and neural and behavioral measures of threat sensitivity. Then, the investigators will conduct a randomized, double-blind, placebo-controlled, between-subjects study to examine the effects of acute inflammation on neural and behavioral measures of threat sensitivity.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a disabling chronic psychiatric disorder that affects more than 8% of the population. New treatments for PTSD symptoms are desperately needed because current pharmacologic and behavioral treatments for PTSD are inadequate or they have low uptake. Accumulating evidence supports elevated inflammation as a new potential treatment target for PTSD. Inflammation is increased in PTSD, and can promote threat sensitivity, a core mechanism underlying several PTSD symptoms. Two major gaps in knowledge prevent progress towards effective anti- inflammatory treatments for PTSD symptoms. First, researchers know little about the relationship between chronic inflammation and exaggerated threat sensitivity. Second, no studies have directly examined the effects of acute inflammation on neural and behavioral measures of threat sensitivity in PTSD. The objective of this study is to uncover the effects of chronic and acute inflammation on neural mechanisms and behavioral measures of threat sensitivity in individuals with and without PTSD symptoms. The central hypothesis is that both chronic and acute inflammation will be associated with exaggerated threat sensitivity overall, with particularly strong relationships in PTSD. The scientific rationale is that establishing a link between elevated inflammation and threat sensitivity in both observational and experimental studies in individuals with and without PTSD symptoms will drive progress towards a targeted approach to identifying effective anti- inflammatory treatments for PTSD symptoms. In particular, this work has the potential to identify a target for clinical trials of anti-inflammatory interventions in PTSD. Guided by preliminary data, hypotheses will be tested by pursuing two specific aims: 1) Examine the association of chronic inflammation with threat sensitivity; and 2) Determine the effects of an acute inflammatory challenge on threat sensitivity. To achieve these aims, 40 participants with moderate to severe PTSD symptoms and 40 age- and body mass index-matched trauma-exposed participants with no history of PTSD will be recruited. The investigators will assess chronic resting levels of inflammation (Aim 1) and will randomize participants to placebo or inflammatory challenge using polysaccharide typhoid vaccine (i.e., endotoxin) (Aim 2) and will use validated functional MRI paradigms and behavioral tasks to assess threat sensitivity.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Veterans aged 30-60.

PTSD Subjects:

* Positive for current chronic moderate to severe PTSD symptoms of at least three months duration as indexed by the Clinically Administered PTSD Scale for DSM 5 (CAPS-5).

Control Subjects:

* Negative for lifetime PTSD.
* Negative for lifetime diagnosis of Mood Disorders, Generalized Anxiety Disorder, Obsessive-Compulsive Disorder and Panic Disorder.

Exclusion Criteria:

All Subjects:

* Lifetime history of any psychiatric disorder with psychotic features, bipolar disorder, panic disorder, obsessive-compulsive disorder, alcohol or substance dependence, or a history of alcohol or substance abuse within the past 2 years.
* Currently exposed to recurrent trauma or have been exposed to a traumatic event within the past 3 months.
* Diagnosis of neurologic disorder, systemic illness affecting central nervous system function, and/or anemia.
* Prominent suicidal or homicidal ideation.
* Current and planned ongoing use of medications that impact inflammation or immune function, or use of such medications in the past 6 months.
* Subjects currently receiving serotonin reuptake inhibitors (SSRIs), benzodiazepine or benzodiazepine receptor agonists, anticonvulsants, atypical antipsychotic medication, any antidepressant medication including trazodone.
* Termination of SSRIs, benzodiazepine or benzodiazepine receptor agonists, anticonvulsants, atypical antipsychotic medication, any antidepressant medication including trazodone in the last month or plans to start these medications during the course of the study.
* Contraindications to Magnetic Resonance Imaging (MRI), which include claustrophobia severe enough to prevent MRI examination and presence of ferrometallic objects in the body that would interfere with MR examination and/or cause a safety risk (e.g., pace makers, implanted stimulators, pumps).
* Contraindications to typhoid vaccine, which include acute febrile illness within the past two weeks, disorders characterized by a deficiency in ability to mount a humoral or cell-mediated immune response, use of anti-malarial medications in past six months, antibiotics in past three months, a history of hypersensitivity to typhoid vaccine or any other vaccine, previous immunization with whole-cell typhoid or live, oral typhoid vaccine, vaccination with the polysaccharide version of the typhoid vaccine within the past 3 year, coagulation disorders and thrombocytopenia.
* Conditions or use of substances that may be associated with inflammation independent of trauma and PTSD, including chronic physical disease.
* History of neurologic disorders, traumatic brain injury (TBI), brain tumor, brain hemorrhage, or head injury with loss of consciousness.
* Women who are currently, or are planning to become, pregnant during the study.

The investigators will not exclude PTSD patients who are receiving psychotherapy, but will apply the following criteria: patients must have been in treatment for 6 months, meet symptomatic criteria for inclusion, and do not have plans to discontinue treatment during the course of the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Neural activity to threat as assessed with functional magnetic resonance imaging | Change from Visit 1 (baseline) to Visit 2 (within two weeks of baseline)
  On visits 1 (baseline) and 2 (post-vaccine or post-placebo administration), participants will perform computerized threat and reward tasks and investigators will measure and compare neural activity between groups (PTSD vs. control) and condition (endotoxin vs. placebo).

SECONDARY OUTCOMES:
Threat sensitivity | Change from Visit 1 (baseline) to Visit 2 (within two weeks of baseline)
  Participants will perform computerized tasks designed to assess threat sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Aoife S O'Donovan, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No